CLINICAL TRIAL: NCT05439018
Title: Effect of Integrated Neuromuscular Inhibition Technique on Subjects with Neck Pain and Forward Head Posture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Somaya Nady Mohamed Elsayed, Assistant lecturer of physical Therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INMI on neck pain and FHP
Record Dates: First submitted 2022-06-23; First posted 2022-06-30 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Neck Pain and Forward Head Posture
Keywords: neck pain; Forward head posture
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: this trial has two groups ,one experimental and one control
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Integrated Neuromuscular Inhibition (Experimental): Integrated Neuromuscular Inhibition in addition to traditional treatment will be received three times a week for eight weeks. Integrated Neuromuscular Inhibition will be contain three combined manual treatment ( ischemic compression , strain counter strain , Muscle energy technique )
  Interventions: Other: Integrated Neuromuscular inhibition
- traditional treatment (Active Comparator): traditional treatment will be received three times a week for eight weeks . traditional treatment in Form of stretching and strenghthening of cervical muscles and postural advices
  Interventions: Other: traditional treatment

INTERVENTIONS:
Other: Integrated Neuromuscular inhibition — Integrated Neuromuscular Inhibition in addition to traditional treatment will be received three times a week for eight weeks. Integrated Neuromuscular Inhibition will be contain three combined manual treatment ( ischemic compression , strain counter strain , Muscle energy technique ) traditional treatment will be received three times a week for eight weeks . traditional treatment in Form of stretching and strenghthening of cervical muscles and postural advices
  Other Names: INMI
  Arms: Integrated Neuromuscular Inhibition
Other: traditional treatment — traditional treatment will be received three times a week for eight weeks . traditional treatment in Form of stretching and strenghthening of cervical muscles and postural advices
  Arms: traditional treatment

SUMMARY:
1. To investigate the effects of integrated neuromuscular inhibition technique for upper trapezius and suboccipital muscles on craniovertebral angle in neck pain and forward head posture subjects.
2. To investigate the effects of integrated neuromuscular inhibition technique for upper trapezius and suboccipital muscles cervical pain intensity level in neck pain and forward head posture subjects.
3. To investigate the effects of integrated neuromuscular inhibition technique for upper trapezius and suboccipital muscles on cervical range of motion in neck pain and forward head posture subjects.
4. To investigate the effects of integrated neuromuscular inhibition technique for upper trapezius and suboccipital muscles on cervical proprioception in neck pain and forward head posture subjects.
5. To investigate the effects of integrated neuromuscular inhibition technique for upper trapezius and suboccipital muscles cervical function in neck pain and forward head posture subjects.

DETAILED DESCRIPTION:
Forward head posture (FHP) is one of the most common types of postural abnormality, and it is generally described as an anterior position of the head in relation to the vertical line of the body's center of gravity. Many researchers have reported that several factors, including headache, neck pain, and musculoskeletal disorders such as temporomandibular disorders or rounded shoulders, are related to FHP . It is associated with shortening of the upper trapezius, the posterior cervical extensor muscles, the sternocleidomastoid muscle and the levator scapulae muscle Forward head posture (FHP) is a forward inclination of the head with cervical spine hyperextension and is associated with shortening of the upper trapezius, the splenius and semispinalis capitis and crevice's, the cervical erector spinae and the levator scapulae musculature . A significant number of the population experiences neck related musculoskeletal problems caused by abnormal forward head posture. Forward Head Posture (FHP) is a common postural deviation reported in the literature, and has been considered as a risk factor for the development of neck pain. Around 61.3% adults with neck pain, working using computers were reported to have FHP In addition, patients with chronic neck pain demonstrated weakness in their deep neck flexors and presented with FHP when distracted. Neck pain is a common disorder characterized by pain, discomfort or soreness experienced in a region between the inferior margin of the occipital bone and T1. Prevalence of neck pain in employees is not the same all over the world. In western countries it has been reported to be between 34% and 54%.As neck pain could become a chronic and disabling symptom, discovering and controlling risk factors seems to be a reasonable prevention strategy. Improper posture could be improved by education and proper reminders to decrease the prevalence of neck pain and increase the quality of life. It is thought that adolescents or patients with neck pain (NP) have a more forward head posture, thus a smaller craniovertebral (CV) angle than age-matched pain-free participants. It was concluded that the CV angle is negatively correlated with the disability of patients with neck pain. So, patients with small CV angle have a greater forward head posture, and the greater the forward head posture, the greater the disability

ELIGIBILITY:
Inclusion Criteria:

1. - Adolescent Female physical therapy students between 18-23 years old
2. BMI between 18.5-25 kg/m²
3. Symptomatic forward head posture with CVA 49° or less.
4. Latent trigger point
5. Neck pain more than 3 months

Exclusion Criteria:

1. Cervical disc
2. Myelopathy or cervical radiculopathy
3. Cervical spine surgery in the past
4. Having received physical therapy in the three months prior to the study
5. Non- rheumatologic diseases as multiple sclerosis, thyroid dysfunction and chronic infection.
6. Rheumatologic condition as poly-articular osteoarthritis, rheumatoid arthritis and advanced cervical spine degenerative diseases. -

Ages: 18 Years to 23 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Craniovertebral angle | up to eight weeks
  Craniovertebral angle (CVA): is the angle formed between a horizontal line through the spinous process of C7 and a line from the tragus of the ear

SECONDARY OUTCOMES:
Neck pain intensity level | up to eight weeks
  Neck pain will measured by visual analogue scale ( VAS) .When responding to a VAS item, patients make marks along 100 mm line at the point they feel represents their current pain state .
  with 100 mm means high level of pain and 0 means no pain
change in Neck Functional disability | up to eight weeks
  Neck disability will measured by English neck disability index (NDI) Questionnaire is composed of a total of 10 questions.Each question has 6 answer options which pertain to a level of severity (0-5) with total score of 50 ,when NDI is high the neck function is the worst
Cervical Range of motion ROM | up to eight weeks
  Cervical Range of motion will measured by clinometer application
Cervical proprioception | up to eight weeks
  Cervical proprioception will measured by clinometer application

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical Therapy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mohamed DA, Kamal RM, Gaber MM, Aneis YM. Combined Effects of Extracorporeal Shockwave Therapy and Integrated Neuromuscular Inhibition on Myofascial Trigger Points of Upper Trapezius: A Randomized Controlled Trial. Ann Rehabil Med. 2021 Aug;45(4):284-293. doi: 10.5535/arm.21018. Epub 2021 Aug 30. PMID 34496471
- [Background] Saadat Z, Hemmati L, Pirouzi S, Ataollahi M, Ali-Mohammadi F. Effects of Integrated Neuromuscular Inhibition Technique on pain threshold and pain intensity in patients with upper trapezius trigger points. J Bodyw Mov Ther. 2018 Oct;22(4):937-940. doi: 10.1016/j.jbmt.2018.01.002. Epub 2018 Jan 17. PMID 30368338